CLINICAL TRIAL: NCT01819168
Title: Antimuscarinic Treatment for Female Patients With Overactive Bladder Syndrome: Comparison of Daytime and Nighttime Dosing
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 102026-E
Record Dates: First submitted 2013-03-21; First posted 2013-03-27 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-02

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this retrospective study is to analyze if nighttime antimuscarincs may be more effective in treating patients with nocturia.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent tolterodine SR treatment once per day for 12 weeks in Department of Obstetrics & Gynecology in National Taiwan University Hospital and Far Eastern Memorial Hospital

Exclusion Criteria:

-

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will perform a retrospective study to review the data of bladder diary, urodynamic studies and clinical data of patients who underwent tolterodine SR treatment once per day for 12 weeks in Department of Obstetrics & Gynecology in National Taiwan University Hospital and Far Eastern Memorial Hospital.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
bladder diary | 3 months
  To clarity any difference of reduction in the episodes of nocturia between these two groups.

SECONDARY OUTCOMES:
Frequency and Urgency | 3 months
  To clarity any difference of reduction in the episodes of urinary frequency and urgency between these two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan